CLINICAL TRIAL: NCT06351020
Title: A Phase III, Open-Label, Multi Center, Randomized Study of LM-302 Versus Treatment of Physician's Choice (TPC) in Patients With CLDN18.2-Positive, Locally Advanced or Metastatic Gastric(GC) and Gastroesophageal Junction(GEJ) Adenocarcinoma.
Brief Title: LM-302 for the Treatment of Subjects With Claudin18.2-Positive Gastric and Gastroesophageal Junction Adenocarcinoma.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LaNova Medicines Zhejiang Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM302-03-101
Record Dates: First submitted 2024-03-15; First posted 2024-04-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced or Metastatic GC and GCJ Adenocarcinoma
MeSH Terms: interventions — apatinib; Irinotecan

STUDY DESIGN:
Intervention Model Description: experimental arm:LM-302 control arm:Apatinib or Irinotecan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-302 (Experimental): Patients will accept LM-302 monotherapy
  Interventions: Drug: LM-302
- Physician's choice Apatinib or Irinotecan (Active Comparator): Patients will accept Apatinib or Irinotecan monotherapy
  Interventions: Drug: Apatinib; Drug: Irinotecan

INTERVENTIONS:
Drug: LM-302 — LM-302 intravenous-injection every 2 weeks on Day 1 of each 14-day cycle
  Arms: LM-302
Drug: Apatinib — The subjects will receive Apatinib orally,qd
  Arms: Physician's choice Apatinib or Irinotecan
Drug: Irinotecan — The subjects will receive Irinotecan intravenous-injection,every 2 weeks on Day 1 of each 14-day cycle
  Arms: Physician's choice Apatinib or Irinotecan

SUMMARY:
This study will assess the efficacy and safety of LM-302 Versus Treatment of Physician's Choice (TPC) in Subjects With locally advanced or metastatic, Claudin (CLDN) 18.2-positive, Gastric or Gastroesophageal Junction Adenocarcinoma who have progressed on or after 2 lines of systemic therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, male and female
* Has histopathologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the gastric/gastroesophageal junction (G/GEJ AC).
* Has received and progressed on at least 2 lines of systemic therapy. A prior (neo)adjuvant systemic therapy that ended within 6 months prior to disease relapse is defined as the first line therapy.
* Centrally confirmed CLDN18.2-positive
* HER2 negative
* At least one measurable lesion according to the solid tumor response Evaluation Criteria (RECIST 1.1)
* ECOG: 0-1
* Expected survival ≥12 weeks;
* Good blood reserve and liver, kidney and coagulation function
* Willing to provide informed consent for study participation.

Exclusion Criteria:

* Within the first 5 years of randomization, there is a history of malignant tumors other than GC/GEJ adenocarcinoma, except for skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ, and skin squamous cell carcinoma that have been cured and cured after treatment
* Individuals with a history of previous immunodeficiency, including those with other acquired or congenital immunodeficiency diseases, or those with a history of organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation
* Urine protein qualitative result ≥ 3+, or urine protein qualitative result is 2+and 24-hour urine protein quantification>1g
* Individuals with a history of severe cardiovascular and cerebrovascular diseases
* Individuals who are unable to control or have serious illnesses, including but not limited to active infections requiring systemic antibiotic treatment within 2 weeks prior to initial medication, interstitial pneumonia/lung disease requiring intervention during screening, and tumor related pain requiring local treatment during screening
* Current peripheral sensory or motor neuropathy ≥ grade 2
* Uncontrollable third space effusion in clinical practice
* Received or planned to undergo major surgery or intervention during the study period within the first 28 days of randomization
* The researcher determined that there are other situations that are not suitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 42 months
  OS was defined defined as the time from date of randomization until death from any cause.
Progression Free Survival (PFS) | up to 42 months
  PFS was defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on Investigator assessment

SECONDARY OUTCOMES:
Objective response rate (ORR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieve a best response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Investigator.
Duration of response (DoR) | Time from initial response (CR or PR) to date of documented disease progression or death (due to any cause) whichever occurs first, up to approximately 42 months
  defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieved CR, PR, or stable disease (SD) for a minimum of 6 weeks during study treatment, based on Investigator assessment.
AE and SAE | From signing the ICF until 28 days after EOT or accept other anti-cancer therapy,up to 40 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0
Evaluate the immunogenicity of LM-302 | up to 42 months
  Anti-drug antibody (ADA) will be detected, the titer of ADA will be evaluated using the validated assay.
Evaluation of pharmacokinetic characteristics of LM-302 | up to 42 months
  Peak Plasma Concentration (Cmax) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of LM-302 | up to 42 months
  Area under the plasma concentration versus time curve (AUC) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of LM-302 | up to 42 months
  Trough concentration will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of total antibody | up to 42 months
  Peak Plasma Concentration (Cmax) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of total antibody | up to 42 months
  Area under the plasma concentration versus time curve (AUC) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of total antibody | up to 42 months
  Trough concentration will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of MMAE | up to 42 months
  Peak Plasma Concentration (Cmax) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of MMAE | up to 42 months
  Area under the plasma concentration versus time curve (AUC) will be evaluated using PopPK model and simulation.
Evaluation of pharmacokinetic characteristics of MMAE | up to 42 months
  Trough concentration will be evaluated using PopPK model and simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, Principal Investigator — Peking Union Medical College Hospital; Jin Li, Principal Investigator — Shanghai East Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality